CLINICAL TRIAL: NCT00463307
Title: Evaluation of Applicability of Urine Based Schistosomiasis Test Strip in the Epidemiologic Mapping and Sampling of Schistosoma Mansoni Infection in Low Endemic Areas of Kenya
Brief Title: Evaluation of the Use of a Urin Test Strip to Determine the Spread of Schistosoma Infections in Areas Where Schistosomiasis Infections Are Low in Kenya
Status: Completed | Type: Observational
Sponsor: DBL -Institute for Health Research and Development (Other)
Other Study IDs: SRP-KY-JK-06
Record Dates: First submitted 2007-04-19; First posted 2007-04-20 (Estimated); Last update posted 2007-10-31 (Estimated); Status verified 2007-10

CONDITIONS: Schistosomiasis Mansoni; Circulating Cathodic Antigen Urine Based Dipstick
Keywords: schistosomiasis; Schistosoma mansoni; Circulating cathodic antigen urine dipstick
MeSH Terms: conditions — Schistosomiasis mansoni; Schistosomiasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate the use of a urine test strip in diagnose schistosoma mansoni in areas of Kenya where the rate of infections are low.

The hypothesis is that the urine strip test is a superior tool to the conventional parasitological tools used to diagnose schistosomiasis mansoni infections in area where there is low transmission

DETAILED DESCRIPTION:
The study will compare the use of the urine test strip with the conventional method used and with a "golden standard" methode, in an area of Kenya where the infection transmission is low. Furthermore will the urine test strip be evaluatied in its ability to monitor the intensity of infections in school children before and after they are been treated for the infections.

A total of 1100 school children in the age between 10 and 18 years will be included in the study. Children have to submitt a stool and a urine sample on three consecutive days. Children who are found to be infected with the schistosomiasis parasite will be offered treatment.

ELIGIBILITY:
Inclusion Criteria:

* Children in the age between 10 and 18 years

Exclusion Criteria:

* Children younger then 10 years of age and children whos parent/guardians did not give informed consents for their participation in the study

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1100 (Actual)
Dates: Start 2006-04; Study Completion 2006-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hussein J Kihara, mr, Principal Investigator — Division of Vector Borne Diseases, Kenya
Locations (1):
- Kenya Medical Research Institute, Nairobi, Kenya